CLINICAL TRIAL: NCT05888064
Title: A Technical Framework for Combining Multi-parametric Imaging With Advanced Modelling in Personalized Radiotherapy
Brief Title: Multi-parametric Imaging in Personalized Radiotherapy
Status: Recruiting | Type: Observational
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Collaborators: Dept. of Electronics, Informatics, Bioengineering, Politecnico di Milano, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: CNAO 43 2021
Record Dates: First submitted 2023-03-03; First posted 2023-06-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Skull Base Chordoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective non-invasive MRI acquisitions are planned to be performed: Prospective non-invasive MRI acquisitions are planned to be performed
  Interventions: Diagnostic Test: diffusion MRI sequences
- retrospective group: patients treated for skull base chordoma with particle therapy

INTERVENTIONS:
Diagnostic Test: diffusion MRI sequences — Diffusion MRI sequences will be optimized to derive more accurate estimates of microstructure and microvasculature of tumour and healthy organs: multiple b-values will be acquired and advanced diffusivity models considered. MRI sequences to derive tumour hypoxia (i.e. indicative of radioresistance) will be also considered along with MR spectroscopy to evaluate tumour microenvironment.
  Groups: Prospective non-invasive MRI acquisitions are planned to be performed

SUMMARY:
The study consists in the retrospective and prospective collection of imaging data (along with clinical information related to treatment) of skull-base chordoma patients treated with particle therapy, to derive imaging biomarkers which, integrated with advanced mathematical models, will allow predicting treatment outcome on a multi-scale basis.

DETAILED DESCRIPTION:
The study design consists of the retrospective collection of routinely-acquired data (CT, MRI and dose maps, along with relevant clinical information) and the prospective acquisition of optimized non-invasive MR imaging data, of skull-based chordoma patients treated with particle therapy (PT) at the National Center for Oncological Hadrontherapy (CNAO, Pavia, Italy).

This data will be stored in a proper repository under CNAO's control, shared with Politecnico di Milano through encrypted channels, and it will be used to implement mathematical models able to predict treatment outcome at different scales (macroscopic, microscopic and radiobiological).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of chordoma of the skull base
* Particle therapy with curative intent
* Karnofsky Performance status greater than or equal to 60
* Patients with macroscopic disease detectable at pre-radiotherapy imaging
* Patients undergoing PT with standardized treatment procedures
* Patients who have signed the written informed consent for research

Exclusion Criteria:

* Metastatic disease
* Palliative treatment
* Other malignancies with disease-free interval < 5 years (excepting pre- cancerous lesions)
* Pregnancy
* Simultaneous CHT or Immunotherapy
* Extensive metal instrumentation/implants
* Patients with autoimmune diseases (ADs) -including collagen-vascular (CVD) and inflammatory bowel (IBD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: skull-based chordoma patients treated with particle therapy at the National Center for Oncological Hadrontherapy (CNAO, Pavia, Italy).
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-08-18 (Estimated)

PRIMARY OUTCOMES:
collect data from MRI acquisition | 1 year from the treatment provided in routine clinical setting
  The prospective part of the study aims to collect data from MRI acquisition. It is not focused on patients treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Iannalfi, MD, Principal Investigator — CNAO National Center of Oncological Hadrontherapy
Locations (1):
- CNAO, Pavia, Pv, Italy